CLINICAL TRIAL: NCT01880021
Title: Characterization of Explanted Hernia Meshes From Human Subjects: A Prospective Study
Brief Title: Synthetic Mesh Explant Study
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 2010-12735
Record Dates: First submitted 2013-05-31; First posted 2013-06-18 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Herniorrhaphy; Humans; Polypropylene; Polytetrafluoroethylene; Histology; Materials Testing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether synthetic hernia mesh materials undergo physical and/or chemical changes while in the body.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 yrs
* Previous placement of hernia mesh material
* Current need for excision of previous mesh placement or Current need for intra-abdominal surgical procedure

Exclusion criteria:

* Age < 18 yrs
* No retained mesh prosthetic.
* Non surgical candidate
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from study investigators' patient population.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2008-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Fibrosis level of explanted mesh | Within 2 weeks
  Each specimen will be graded and given fibrosis score of 0 - 4 to establish the degree of inflammation/foreign body reaction that occurred while mesh was in vivo.

SECONDARY OUTCOMES:
Tensile strength of explanted mesh | Within 2 weeks
  Each specimen will be tested for tensile strength to determine force versus displacement.
Collagen protein levels of explanted mesh. | Within 2 weeks
  The total amount of collagen and non-collagenous proteins in cultured cell layers and tissue sections by differential staining with two dyes, sirius red and fast green. Sirius Red binds to all types of collagen, whereas fast green stains non-collagenous proteins.
Number of subjects with history of radiation to abdomen/pelvis | Within 2 weeks
  Identify possible clinical characteristics which affect mesh degradation.
Number of subjects with history of chemotherapy | Within 2 weeks
  Identify possible clinical characteristics which affect mesh degradation.
Number of subjects with corticosteroid/immunosuppression therapy | Within 2 weeks
  Identify possible clinical characteristics which affect mesh degradation.
Number of subjects with history of tobacco use | Within 2 weeks
  Identify possible clinical characteristics which affect mesh degradation.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Brunt, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States